CLINICAL TRIAL: NCT00186862
Title: Phase I Study of Chemokine and Cytokine Gene Modified Allogeneic Neuroblastoma Cells For Treatment of Relapsed/Refractory Neuroblastoma Using a Retroviral Vector
Brief Title: Gene Modified Allogeneic Neuroblastoma Cells For Treatment of Relapsed/Refractory Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Texas Children's Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Gregory Hale, MD, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYCHAL
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Immunotherapy; Gene therapy
MeSH Terms: conditions — Neuroblastoma | interventions — Interleukin-2; Immunotherapy; Genetic Engineering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — A genetically modified (retroviral) allogeneic tumor vaccine coupled with the human interleukin-2. Patients were treated with 4 injections of these gene-modified tumor cells. The first two were given at weeks 1 and 2. Patients then had a 2 week rest and the remaining 2 injections were given at weeks 4 and 5. A complete evaluation for evidence of toxicity and response were performed at week 8.
  At this week 8 evaluation, if there was no excessive toxicity, progressive disease requiring therapy, and if more transduced cells are available, patients had the option to receive 4 additional injections. These additional injections were separated by 1 month at the higher of the two dosage levels originally received.
  Other Names: Immunotherapy; gene transfer

SUMMARY:
Neuroblastoma affects approximately 500 children a year in the United States. When the tumor occurs in infants, it is frequently localized and responds well to therapy. Even disseminated disease can be eradicated in about 75% of infants, and indeed may undergo spontaneous remission. In older children, the prognosis is far worse, and 80% or more of those with disseminated tumor can be expected to relapse within 3 years.

This study will utilize the concept of exploiting the immune system to eradicate neuroblastoma. In tumors in which there is consistent expression of tumor specific antigens as part of the malignant process, it may be possible to generate immune T-cells ex-vivo or in-vivo by using the specific protein or peptide(s) derived therefrom and eradicate the tumor. This study will evaluate the use of four to eight injections of IL-2 gene-transduced autologous neuroblastoma cells to induce a local, polyclonal T-cell infiltrate as well as an anti-tumor immune response.

DETAILED DESCRIPTION:
Secondary objectives for this protocol included the following:

* To determine whether major histocompatibility complex (MHC) restricted or unrestricted antitumor immune responses are induced by injection of modified allogeneic neuroblasts and the cell doses required to produce these effects.
* To obtain preliminary data on the antitumor effects of this treatment regimen.

ELIGIBILITY:
* Diagnosis of recurrent advanced stage neuroblastoma.
* Must have a life expectancy of at least 8 weeks.
* Must have recovered from the toxic effects of all prior chemotherapy before entering this study, and have an absolute neutrophil count of >500/mm3.
* Not be currently receiving any investigational agents or have not received any tumor vaccines within the previous six months.
* Bilirubin <1.5 mg/dl.
* Creatinine <1.5 mg/dl.
* ECOG performance status of 0-2 as below:
* Does not have rapidly progressive disease.
* Not pregnant or lactating.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 1998-08; Primary Completion 2000-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
• To determine the safety of up to eight subcutaneous injections of allogeneic neuroblastoma cells that have been genetically modified by retroviral vectors to secrete lymphotactin and Interleukin-2 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Hale, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org